CLINICAL TRIAL: NCT02427204
Title: Outcomes in Liver Disease Patient With and Without HIV Co-infection-Sub Study 2: HCV Treatment: Health Related Quality of Life, Fatigue, Work Productivity, Liver Status and Cost-per-SVR/Health Care Utilization
Brief Title: Outcomes in Liver Disease Patient With and Without HIV Co-infection-Sub Study 2: HCV Treatment: Health Related Quality
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1959
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Infection
Keywords: Hepatitis C infection; Hepatitis C treatment
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main questions being addressed are (1) how patient reported outcomes change during treatment for HCV, (2) how treatment impacts liver function and liver status, and (3) how much treatment costs from the payer's perspective and the patient's perspective. The hypothesis being tested is that treatment has a negative effect on the quality of life during treatment. The negative effect is expected to be temporary. Successful treatment, which is equated with a virological cure of the infection, is expected to result in an improvement in quality of life compared to baseline and to improvement in markers of liver function and liver status. Costs of treatment are expected to be $80,000-$200,000 per virological cure.

DETAILED DESCRIPTION:
The objectives of the study are to collect information about patient reported outcomes before, during, and after treatment for hepatitis C virus infection, to determine the impact of treatment on liver function and stiffness (an indicator of inflammation and fibrosis), and to determine the cost of treatment.

The main questions being addressed are (1) how patient reported outcomes change during treatment for HCV, (2) how treatment impacts liver function and liver status, and (3) how much treatment costs from the payer's perspective and the patient's perspective. The hypothesis being tested is that treatment has a negative effect on the quality of life during treatment. The negative effect is expected to be temporary. Successful treatment, which is equated with a virological cure of the infection, is expected to result in an improvement in quality of life compared to baseline and to improvement in markers of liver function and liver status. Costs of treatment are expected to be $80,000-$200,000 per virological cure.

The purpose of the study is to give patients and providers information about what to expect while undergoing treatment for HCV and to provide information for future cost-effectiveness studies. Previous studies of liver biopsy and transient elastography demonstrate that liver scarring regresses in a significant percentage of patients who achieve an SVR; however, the majority of patients who had liver cirrhosis at the time they achieved an SVR continued to have portal hepatitis and high levels of alpha smooth muscle actin ( D'Ambrosio R, et al., Hepatology, 2012). Particularly because interferon is known to cause autoimmune disease, it is possible that some residual liver abnormalities are due to interferon exposure. If this is the case, liver abnormalities may regress more rapidly and completely in patients receiving interferon-free regimens. Currently, there are no real-world data about the impact of new regimens on liver status as measured by transient elastography. This project will fill an important gap by providing information about changes in liver stiffness in patients receiving the newest therapies for HCV.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Positive test for HCV RNA and planning to start HCV treatment soon
* Able to travel to Mount Sinai
* Must understand and speak English
* Planning to initiate treatment for HCV infection in the near future
* Willing to sign informed consent and participate

Exclusion Criteria:

* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients initiating treatment for HCV infection are the source of potential subjects.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-06; Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

PRIMARY OUTCOMES:
Change in vitality score, Short form 36 (SF36) | baseline and week 24
  Change in vitality score at week 24 as compared to baseline

SECONDARY OUTCOMES:
Change in work productivity and activity impairment (WPAI) questionnaire | baseline and week 24
  Change in activity at week 24 as compared to baseline
Change in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | baseline and week 24
  Change in function at week 24 as compared to baseline
Change in quality of life symptoms, Chronic Liver Disease Questionnaire-HCV (CLDQ-HCV) | baseline and week 24
  Change in quality of life symptoms at week 24 as compared to baseline
Change in Medication adherence survey | baseline and week 24
  Change in medication adherence at week 24 as compared to baseline
Change in Medication and co-morbidities questionnaire | baseline and week 24
  Change in medication and co-morbidities at week 24 as compared to baseline
Lost wages: Change in work ability | baseline and week 24
  Change in work ability at week 24 as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrea D Branch, PhD, Principal Investigator — Icahn School of Medicine
Locations (1):
- Icahn School of Medicine, New York, New York, United States